CLINICAL TRIAL: NCT03299517
Title: PROSPECTIVE ANALYSIS BETWEEN AMIODARONE Versus LIDOCAINE IN PATIENTS WITH STABLE VENTRICULAR TACHYCARDIA IN THE EMERGENCY ROOM
Brief Title: PROSPECTIVE ANALYSIS BETWEEN AMIODARONE Versus LIDOCAINE IN SVT
Acronym: AMIOLIDO-VT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PSInCor-AMIOLIDO-VT
Record Dates: First submitted 2017-09-27; First posted 2017-10-03 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Arrhythmias Ventricular
Keywords: lidocaine; amiodarone
MeSH Terms: interventions — Lidocaine; Anti-Arrhythmia Agents; Amiodarone

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine (Experimental): Initial dose: antiarrythmic drugs Lidocaine (1.5 mg / kg EV in 30 minutes).
  Adittional dose: Lidocaine (0.75 mg / kg EV in 30 minutes).
  Interventions: Drug: Antiarrythmic Drugs
- amiodarone (Experimental): Initial dose: antiarrythmic drugs Amiodarone (5 mg / kg EV in 30 minutes)
  Adittional dose: Amiodarone (3 mg / kg EV in 30 minutes)
  Interventions: Drug: Antiarrhythmic drugs

INTERVENTIONS:
Drug: Antiarrythmic Drugs — Patient will be randomly randomized 1: 1 for the antiarrythmic drugs. If there is no reversal and there is no adverse event, a further dose of the same pre-administered medicinal product will be performed in another 30 minutes.
  Other Names: lidocaine
  Arms: lidocaine
Drug: Antiarrhythmic drugs — Patient will be randomly randomized 1: 1 for the the antiarrythmic drugs. If there is no reversal and there is no adverse event, a further dose of the same pre-administered medicinal product will be performed in another 30 minutes.
  Other Names: amiodarone
  Arms: amiodarone

SUMMARY:
Introduction: Recent studies have suggested that other medications may be superior to amiodarone in controlling ventricular arrhythmias. However, a prospective and randomized comparison with lidocaine has not yet been described.

Objective: This study aims to evaluate the effectiveness and safety of the use of amiodarone versus lidocaine in patients with stable ventricular tachycardias.

Methodology: For this, a unicentric, randomized and prospective study will be carried out, in which the two drugs will be administered in a comparative manner. Hospital data (test results, medical outcomes, arrhythmia reversal, complications) of patients will be analyzed for safety and effectiveness.

Expected results: The use of lidocaine is not inferior to amiodarone in the tolerability and reversion of stable ventricular tachycardias.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women> 18 years old
* Presence of sustained ventricular tachycardia with HR> 120 bpm
* Systolic blood pressure> 90 mmHg
* No signs of poor peripheral perfusion
* Absence of dyspnea
* Absence of severe angina
* Signed consent form

Exclusion Criteria:

* Pregnancy
* Hemodynamic instability
* Body mass index greater than 40 kg / m2
* Use of intravenous amiodarone or lidocaine in the last 24 hours
* Acute coronary syndrome
* Presence of tachycardia with irregular or supraventricular RR
* Contraindications to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2019-08-02 (Estimated); Study Completion 2022-08-02 (Estimated)

PRIMARY OUTCOMES:
Signs of peripheral hypoperfusion and shock | 1 hour
  hypoperfusion and shock
Signs of pulmonary congestion | 1 hour
  dyspnea, orthopnea, onset of pulmonary rales or drop in oximetry.
Severe hypotension | 1 hour
  systolic blood pressure <70 mmHg if the previous one is <100 mmHg or systolic blood pressure <80 mmHg if the previous one is > 100 mmHg).
HR increase | 1 hour
  HR increase> 20 bpm.
The appearance of polymorphic TV. | 1 hour
  polymorphic TV.
Lowering the level of consciousness. | 1 hour
  glasgow < 15

SECONDARY OUTCOMES:
effectiveness of reversal | 1 hour
  sinusal rhythm
time required for reversal | 1 hour
  sinusal rhythm

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Soeiro, MD, Principal Investigator — Unidade Clínica de Emergência
Locations (1):
- Instituto do Coração - HMFMUSP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Somberg JC, Bailin SJ, Haffajee CI, Paladino WP, Kerin NZ, Bridges D, Timar S, Molnar J; Amio-Aqueous Investigators. Intravenous lidocaine versus intravenous amiodarone (in a new aqueous formulation) for incessant ventricular tachycardia. Am J Cardiol. 2002 Oct 15;90(8):853-9. doi: 10.1016/s0002-9149(02)02707-8. PMID 12372573
- [Result] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995